CLINICAL TRIAL: NCT06720090
Title: Light Therapy for Obsessive-compulsive Disorder: A Circadian Medicine Approach
Brief Title: Light Therapy for Obsessive-compulsive Disorder (OCD)
Acronym: KLTO
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rebecca C. Cox, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH137376 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-12-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-03

CONDITIONS: OCD
Keywords: ocd; sleep; light therapy; circadian; behavioral treatment
MeSH Terms: conditions — Compulsive Personality Disorder | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Higher dose (Experimental): Participants will be given wearable light therapy devices that emit a higher light intensity.
  Interventions: Behavioral: Light therapy
- Lower dose (Sham Comparator): Participants will be given wearable light therapy devices that emit a lower light intensity.
  Interventions: Behavioral: Light therapy

INTERVENTIONS:
Behavioral: Light therapy — 5 weeks of light therapy administered via wearable light therapy glasses worn for 1 hour each morning after awakening.

SUMMARY:
The goal of this clinical trial is to test whether light therapy is effective for reducing symptoms in young adults with OCD and late bedtimes (1am or later). The main question[s] it aims to answer are:

Does light therapy reduce OCD symptoms? Does light therapy advance the circadian clock? If there is a comparison group: Researchers will compare a higher dose of light therapy to a lower dose to see if dose amount affects symptom reduction.

Participants will asked to:

1. Wear light therapy glasses for 1 hour each morning and complete a daily light therapy log for 5 weeks
2. Track their sleep every day with a wearable monitor and an electronic sleep diary for 5 weeks
3. Complete a 1-time assessment of sensitivity to light exposure
4. Complete self-report measures of OCD 4 times/day at baseline (2 weeks), mid-treatment (1 week), and end of treatment (1 week)

ELIGIBILITY:
Inclusion Criteria:

1. Primary DSM-5 OCD diagnosis
2. Bedtime 0100 or later
3. Age 18-35
4. English speaking

Exclusion Criteria:

1. Subjects must not be currently participating in another research study that would influence their participation in our study.
2. Diagnostic status
3. Treatment status
4. Night shift work or travel more than 1 time zone outside of Central Standard Time (CST) in the past month
5. Pregnancy status
6. Medication status
7. Regular nicotine or marijuana use

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive-Compulsive Scale (YBOCS) | Administered at baseline, in treatment week 3, and post-treatment (3 administrations over 7 weeks)
  A retrospective clinical interview of OCD symptom severity. Score range from 0 to 40 and higher scores indicate more severe OCD symptoms.
Daily Perseverative Thinking Questionnaire | Administered 4 times/day for 2 weeks at baseline, 4 times/day for 1 week in treatment week 3, and 4 times/day for 1 week in treatment week 5
  Self-report measure of momentary transdiagnostic repetitive negative thinking. Score range from 6 to 42 and higher scores indicate more severe repetitive negative thinking.

SECONDARY OUTCOMES:
Circadian melatonin phase | At baseline and post-treatment (after 5 weeks of treament)
  Dim light melatonin onset assessed by taking hourly saliva samples in dim light conditions for 10 hours beginning 7 hours before typical bedtime and ending 2 hours after typical bedtime.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cox, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes